CLINICAL TRIAL: NCT00005390
Title: Family Process, Adherence, and Child Asthma Outcome
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4296; R01HL053391 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To examine the role of family processes in asthma regulation in three groups of children with mild to moderate asthma.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The study, which was ancillary to the Childhood Asthma Management Program (CAMP), clarified the extent to which and the mechanisms whereby specific family processes might be protective or deleterious in the adherence behaviors and treatment outcome in three groups of children with mild to moderate asthma: 80 children participating in the Denver site of the CAMP, 80 children receiving asthma-related care in a large, nationally recognized health maintenance organization, and 60 children recruited by using school records to identify children with asthma receiving their care in a variety of different health care systems across the Denver metropolitan area. The study examined the extent to which family process variables were cross-sectionally associated with and longitudinally influenced adherence to asthma treatment and asthma treatment outcome as well as the consistency of this relationship across the three sites. The study also determined whether adherence with treatment mediated the relationship between specific family processes and asthma treatment outcome, as well as the consistency of this relationship across the three sites.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-08; Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Wamboldt — National Jewish Center for Immunology & Respiratory Medicine

REFERENCES:
- [Background] Cohen SY, Wamboldt FS. The parent-physician relationship in pediatric asthma care. J Pediatr Psychol. 2000 Mar;25(2):69-77. doi: 10.1093/jpepsy/25.2.69. PMID 10820945
- [Background] Wamboldt FS, Spahn JD, Klinnert MD, Wamboldt MZ, Gavin LA, Szefler SJ, Leung DY. Clinical outcomes of steroid-insensitive asthma. Ann Allergy Asthma Immunol. 1999 Jul;83(1):55-60. doi: 10.1016/S1081-1206(10)63513-2. PMID 10437817
- [Background] Gavin LA, Wamboldt MZ, Sorokin N, Levy SY, Wamboldt FS. Treatment alliance and its association with family functioning, adherence, and medical outcome in adolescents with severe, chronic asthma. J Pediatr Psychol. 1999 Aug;24(4):355-65. doi: 10.1093/jpepsy/24.4.355. PMID 10431501
- [Background] Gabriels RL, Wamboldt MZ, McCormick DR, Adams TL, McTaggart SR. Children's illness drawings and asthma symptom awareness. J Asthma. 2000;37(7):565-74. doi: 10.3109/02770900009090811. PMID 11059523
- [Background] Wamboldt MZ, Wamboldt FS. Role of the family in the onset and outcome of childhood disorders: selected research findings. J Am Acad Child Adolesc Psychiatry. 2000 Oct;39(10):1212-9. doi: 10.1097/00004583-200010000-00006. PMID 11026173
- [Background] Wamboldt FS, Bender BG, O'Connor SL, Gavin LA, Wamboldt MZ, Milgrom H, Szefler SJ, Ikle D, Rand C. Reliability of the model MC-311 MDI chronolog. J Allergy Clin Immunol. 1999 Jul;104(1):53-7. doi: 10.1016/s0091-6749(99)70113-2. PMID 10400839
- [Background] Frankel K, Wamboldt MZ. Chronic childhood illness and maternal mental health--why should we care? J Asthma. 1998;35(8):621-30. doi: 10.3109/02770909809048964. PMID 9860082
- [Background] Wamboldt MZ, Schmitz S, Mrazek D. Genetic association between atopy and behavioral symptoms in middle childhood. J Child Psychol Psychiatry. 1998 Oct;39(7):1007-16. PMID 9804033
- [Background] Wamboldt MZ, Fritz G, Mansell A, McQuaid EL, Klein RB. Relationship of asthma severity and psychological problems in children. J Am Acad Child Adolesc Psychiatry. 1998 Sep;37(9):943-50. doi: 10.1097/00004583-199809000-00014. PMID 9735613
- [Background] Wamboldt MZ, Wamboldt FS, Gavin L, McTaggart AS. A parent-child relationship scale derived from the child and adolescent psychiatric assessment (CAPA). J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):945-53. doi: 10.1097/00004583-200108000-00017. PMID 11501695
- [Background] Wenzel SE, Morgan K, Griffin R, Stanford R, Edwards L, Wamboldt FS, Rogenes P. Improvement in health care utilization and pulmonary function with fluticasone propionate in patients with steroid-dependent asthma at a National Asthma Referral Center. J Asthma. 2001 Aug;38(5):405-12. doi: 10.1081/jas-100001495. PMID 11515977
- [Background] Millikan E, Wamboldt MZ, Bihun JT. Perceptions of the family, personality characteristics, and adolescent internalizing symptoms. J Am Acad Child Adolesc Psychiatry. 2002 Dec;41(12):1486-94. doi: 10.1097/00004583-200212000-00021. PMID 12447036
- [Background] Ho J, Bender BG, Gavin LA, O'Connor SL, Wamboldt MZ, Wamboldt FS. Relations among asthma knowledge, treatment adherence, and outcome. J Allergy Clin Immunol. 2003 Mar;111(3):498-502. doi: 10.1067/mai.2003.160. PMID 12642828
- [Background] Fiese BH, Wamboldt FS. Tales of pediatric asthma management: family-based strategies related to medical adherence and health care utilization. J Pediatr. 2003 Oct;143(4):457-62. doi: 10.1067/S0022-3476(03)00448-7. PMID 14571219